CLINICAL TRIAL: NCT05807360
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "Hyaluronic Acid (HA)-Based Eyedrops" Used to Relieve Dry Eye Symptoms.
Brief Title: PMCF Study to Evaluate Performance and Safety of "Hyaluronic Acid (HA)-Based Eyedrops" Used to Relieve Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R1-HA
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye; Dry Eye Disease; Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Hyaluronic acid eye drops

INTERVENTIONS:
Device: Hyaluronic acid eye drops — Hyaluronic acid (HA)-based eyedrops

SUMMARY:
Dry eye disease (DED), also called keratoconjunctivitis sicca, is a common ocular condition characterized by a loss of homeostasis of the tear film and inflammation of the ocular surface. The typical symptoms of DED include irritation, discomfort, blurred or fluctuating vision.

Over the counter (OTC) artificial tears are typically the first line of dry eye treatment; they are meant to supplement the tears that cover the eye's surface. OTC products mimic the different layers of the tear film in order to maintain ocular hydration.

HA is found in higher concentrations in the vitreous humor of the eye, cartilage, and the synovial fluid. As a component of the tear film, HA increases the viscosity of the tear film and hydrates and lubricates the ocular surface. HA possesses intrinsic water retention properties, viscoelasticity, and favors the healing of corneal and conjunctival epithelium.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "HA-based eyedrops" used as intended to relieve dry eye symptoms.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of "HA-based eyedrops" according to the IFU.

"Hyaluronic Acid (HA)-based eyedrops" are medical devices used as intended to improve the discomfort due to dry eye (for intrinsic and/or extrinsic causes), contact lenses wearing and/or eye surgery.

Each Subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), one of the "Hyaluronic Acid (HA)-based eyedrops" products can be dispensed to the enrolled Subjects, depending on Investigator clinical evaluation, and severity of the disease.

The patient will perform 2 on site visits (V0 and V2/EOS). To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events (AEs) and concomitant medications intake.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* Male & Female Aged ≥ 18 years at the time of the signature of the ICF;
* Patients with ophthalmic discomfort due to dry eye for intrinsic and/or extrinsic causes, contact lenses wearing and/or eye surgery;
* WIlling not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Suspected alcohol or drug abuse;
* Known hypersensitivity or allergy to IP components;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases, diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer Test I: to evaluate the performance of the "HA-based eyedrops" used to relieve dry eye symptoms due to both intrinsic and extrinsic causes, through Schirmer I test | From Baseline (V0 = Day 0) at 1 month (EOS/V2 = Day 30)

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI): to evaluate the performance of the "HA-based eyedrops" used to relieve eye discomfort sensation | From Baseline (V0 = Day 0) at 1 month (EOS/V2 = Day 30)
Change in Tear Break-up Time (TBUT): to evaluate the performance of the "HA-based eyedrops" used to relieve ophthalmic stress due to prolonged use of contact lenses or surface eye surgery, through the TBUT test | From Baseline (V0 = Day 0) at 1 month (EOS/V2 = Day 30)
To evaluate the safety and tolerability of the "HA-based eyedrops" through Visual Analogical Scale (VAS) - evaluation of symptoms related to dry eye disease (burning, fatigue, discomfort, redness) | End of study visit (EOS/V2 = Day 30)
  Visual Analogical Scale Minimum value = 0 Maximum value = 10 Higher scores mean a better outcome
To evaluate the patient satisfaction of the "HA-based eyedrops" through a 5-points Likert Scale | End of study visit (EOS/V2 = Day 30)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico "G.Rodolico - San Marco", Catania, CT, Italy